CLINICAL TRIAL: NCT06907784
Title: PHOENIX TRIAL - A PILOT RANDOMISED CONTROLLED TRIAL OF PRE-EMPTIVE PHARMACOGENOMICS IN ACUTE CARE SETTINGS WITH HEALTH ECONOMIC EVALUATIONS
Brief Title: PRE-EMPTIVE PHARMACOGENOMICS IN ACUTE CARE SETTINGS WITH HEALTH ECONOMIC EVALUATIONS (PHOENIX TRIAL)
Acronym: PHOENIX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INGN24MG113
Record Dates: First submitted 2025-03-14; First posted 2025-04-02 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pharmacogenomic Drug Interaction
Keywords: Gene-drug; Gene panel; Polypharmacy; Adverse drug reaction; Health economics; pharmacogenomics
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Pharmacogenomic testing will be performed immediately in the intervention group with any resultant drug change by the treating clinician
  Interventions: Diagnostic Test: Pharmacogenomic testing
- Standard of Care (Other): Pharmacogenomic testing (from the stored buccal swab sample) will be performed only at three months in the standard of care arm group with any resultant drug change by the treating clinician.
  Interventions: Diagnostic Test: Pharmacogenomic testing

INTERVENTIONS:
Diagnostic Test: Pharmacogenomic testing — The PGx testing will analyse genetic variants across 16 key pharmacogenes in each given DNA sample, all of which focus on variants with established implications for drug response as recommended by published Clinical Pharmacogenetics Implementation Consortium (CPIC) and the Dutch Pharmacogenetics Working Group (DPWG) guidelines Testing will be performed immediately in the intervention arm or at three months in the standard of care arm.

SUMMARY:
It is known that individuals respond differently to the same medicine with some people benefitting, some experiencing no effect and others suffering side-effects or even coming to harm. Some of the differences in response to medications can be explained by our genes. Genes are short sections of DNA. Each individual has over 20,000 different genes. Genes carry instructions for making the proteins needed to build things within the body including the sites where medicines act. Pharmacogenomics is the study of how our genes affect the way our body responds to medications.

Doctors can test for gene variations that might put an individual at risk of severe side-effects or mean that they are likely to receive no benefit from a specific medicine. Though not widely available in the NHS, testing allows doctors and patients to chose a different dose or avoid the medicine completely. It is estimated that almost everyone in the population (>95%) carries at least one gene variation that affects our response to medicines.

The PHOENIX study will recruit 4,000 participants who are admitted to hospital or attend an outpatient clinic who require a new drug prescription. The new drug prescription will be one who known pharmacogenomic implications. A cheek (buccal) swab will be taken which can be used to test a large number of genes known to alter the response to medicines. Around half of the participants will be tested immediately whilst the other half will have the test after three months. The results of the test relevant to each patients new prescription will enable the doctor prescribing to determine if any changes to that medicine would be beneficial. Information will be collected about participants quality of life, subsequent admissions to hospital, medication changes and side-effects. An assessment of cost saving to the NHS will also be made.

DETAILED DESCRIPTION:
PHOENIX is a pilot two-group parallel randomised trial aimed at generating preliminary evidence on the effectiveness of a pharmacogenomics (PGx) intervention in reducing adverse drug reactions (ADR) and treatment failures in patients (hospitalised or attending secondary care specialist clinics). Additionally, it will provide early insights into health-economic impact of such PGx-guided care. Pharmacogenomic analysis will be conducted on DNA extracted from buccal swab samples taken at consent. This Trial will be performed according to the UK Policy Framework for Health and Social Care Research (2023).

The trial will recruit adult participants, admitted to wards or attending specialist outpatient clinics in Queen Elizabeth University Hospital (QEUH), Glasgow, where the selected PGx drugs are frequently prescribed: General Medicine (all specialities and receiving areas), Medicine for the Elderly, Cardiology, Stroke, Diabetes and Endocrinology, Infectious Diseases, Rheumatology, Neurology, General Surgery, Vascular Surgery, Urology, ENT and Orthopaedics.

Potential participants will be identified by the prescription of a new medicine with pharmacogenomic implications on the HEPMA electronic prescribing system, trial team visit to ward areas, treating clinician or patients self identifying on inpatient ward areas. Drug caps will be in place throughout the trial to prevent over-recruitment of one or more commonly prescribed medications. Potential participants approached by study team and offered PIS/invite. Potential participants contact study team to opt-in or study team return to ask if interested in study +/- further discussion. Written informed consent will be given by each participant or their legal representative is they are deemed to be lacking capacity.

Maximum Total 4000 Intervention arm: 1000 to 2000 Standard of care arm: 1000 to 2000

All participants will provide a buccal swab (mouth swab) for genetic testing. All samples will have DNA extracted on receipt of the sample. Pharmacogenomic testing will be performed immediately for those in the intervention arm or stored and tested at six month in the standard of care arm.

The pharmacogenomic report will be returned to the clinician with responsibility for the patients care (at baseline for intervention or three months for standard of care) with a recommendation regarding the medicine if changes are suggested. This will unblind the treating clinician and potentially the patient if medication changes are made for the intervention group.

All participants will be asked to complete questionnaires on quality of life (monthly for three months), medication adherence and adverse drug reactions (monthly for three months).

Blood testing will be carried out for safety (usual clinical care) at approximately four weeks, dependent on the index drug.

Further information will be collected through West of Scotland Safe Haven on new medication prescriptions, hospital admissions and deaths. This will require the participants CHI (community health index) number to be linked to their Safe Haven data but data will be returned to the researchers in anonymised form.

ELIGIBILITY:
Inclusion Criteria INPATIENTS Age ≥18 years

* Capable of giving informed consent directly or via a legal representative (e.g., next of kin, welfare guardian, health care power of attorney).
* Participants who are newly prescribed one of the trial-eligible index drugs during their hospital stay may be approached for consent. Consent should be obtained within 3 days of the first dose of the index drug being administered. If there is a clear clinical plan documented on HEPMA indicating that the patient will be started on an eligible drug (but has not yet received the first dose), consent may be obtained in anticipation. However, formal trial enrolment will only occur once the first dose of the index drug has been administered.
* Participant must not have a prescription for this drug in the previous 3 months.
* Participant is able to provide a cheek swab
* Participant is able to take part and be followed-up for at least 12 weeks.
* Participant is resident in NHSGGC health board area OUTPATIENTS
* Age ≥18 years
* Capable of giving informed consent directly or via a legal representative (e.g., next of kin, welfare guardian, health care power of attorney).
* Participants who are expected to be prescribed a trial-eligible drug during their outpatient clinic visit may be approached for consent prior to starting the medication. In these cases, formal trial enrolment will only occur once the patient has confirmed that they have received and started the prescribed medication
* Participant must not have a prescription for this drug in the previous 3 months.
* Participant is able to provide a cheek swab
* Participant is able to take part and be followed-up for at least 12 weeks.
* Participant is resident in NHSGGC health board area.

Exclusion Criteria INPATIENTS

* Inability to give informed consent directly or via a legal representative.
* Non-English speakers without translation support.
* Participants co-enrolled in other trials where a medication is one of the index drug is part of the trial protocol.
* Inability to give informed consent directly or via a legal representative.
* Non-English speakers without translation support.
* Participants co-enrolled in other trials where a medication is one of the index drug is part of the trial protocol.
* Life expectancy estimated to be less than 6 months by treating clinical team.
* Severe illness limiting participation (investigator discretion).
* Duration of index drug total treatment length is planned to be less than seven consecutive days.
* Not registered with a General Practitioner.
* No fixed address.
* Participant is, in the opinion of the Investigator, not suitable to participate in the trial.
* Participant has existing impaired hepatic or renal function for which a lower dose or alternate drug selection is already part of current routine care.
* Estimated glomerular filtration rate greater than 15 ml/min/1.73m2 (except for participants with a renal transplant commenced on tacrolimus, who may be included regardless of eGFR, provided they are not on dialysis).eGFR result obtained at screening or within the last 6 months or patients record confirming history of CKD 5
* Participants on any form of dialysis.
* Participant with advanced liver failure (stage Child-Pugh C).
* Participants with liver transplant.
* Participants with allogeneic haematopoietic stem cell transplant.
* Participants previously enrolled in the PHOENIX trial.
* Participant who has declined participation and has declined reapproach for subsequent drugs.
* Index drug exceeding trial drug cap. OUTPATIENTS
* Inability to give informed consent directly or via a legal representative.
* Non-English speakers without translation support.
* Participants co-enrolled in other trials where a medication is one of the index drug is part of the trial protocol.
* Life expectancy estimated to be less than 6 months by treating clinical team.
* Severe illness limiting participation (investigator discretion).
* Duration of index drug total treatment length is planned to be less than seven consecutive days.
* Not registered with a General Practitioner.
* No fixed address.
* Participant is, in the opinion of the Investigator, not suitable to participate in the trial.
* Participant has existing impaired hepatic or renal function for which a lower dose or alternate drug selection is already part of current routine care.
* Estimated glomerular filtration rate greater than 15 ml/min/1.73m2 (except for participants with a renal transplant commenced on tacrolimus, who may be included regardless of eGFR, provided they are not on dialysis)..eGFR result obtained at screening or within the last 6 months or patients record confirming history of CKD 5.
* Participants on any form of dialysis.
* Participant with advanced liver failure (stage Child-Pugh C).
* Participants with liver transplant.
* Participants with allogeneic haematopoietic stem cell transplant.
* Participants previously enrolled in the PHOENIX trial.
* Participant who has declined participation and has declined reapproach for subsequent drugs.
* Index drug exceeding trial drug cap.

Re-approach Criteria: Previously declined patients will only be re-approached in subsequent admissions six-months after the first approach.

* We wish to ensure that no more than 20% of participants are included on the basis of any single index drug. The numbers recruited on each index drug will be monitored and recruitment on specific drugs may be limited, or paused, at times throughout the study. This process will be administered by the Trial Management group, and monitored by the Trial Steering Committee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite of ADRs and/or treatment failures | 3 months
  Composite of ADRS (CTCAE ≥2) and/or treatment failures (applies to specific drugs where treatment failure is captured by hospital admissions with the condition for which the index drug was commenced).

SECONDARY OUTCOMES:
5-level EQ-5D version (EQ-5D-5L) EuroQol | 3 months
  Assess changes in quality of life using the EQ-5D-5L questionnaire administered monthly over three months to explore the impact of PGx-guided care on participants' overall well-being.
  The EQ-5D-5L questionnaire will comprise of ive dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS
PGx Result Utilisation in Intervention Arm | 3 months
  Measure the proportion of participants in the intervention arm who receive at least one drug/dose selection or modification based on PGx test results, offering insight into clinical application.
PGx Result Utilisation in Standard Care Arm (Post-Delayed Genotyping) | 3 months
  For participants in the standard care arm, determine the proportion who receive at least one drug/dose modification after delayed genotyping, highlighting the potential impact if PGx results were available at baseline.
Frequency of Actionable Genotypes at Baseline | 7 days
  Report the frequency of actionable genotypes that lead to drug/dose selection or modification of all drugs, including the index drug, at baseline.
Frequency of Actionable Genotypes for New Prescriptions During Follow-Up | 7 days - 3 months
  Report frequencies of actionable genotypes that indicate drug/dose selection or modification for any new prescriptions issued between 7 and 90 days post-randomisation.
Ordinal analysis of adverse drug reaction (ADR) severity | 3 months
  Evaluate ADR severity across different grades using NCI-CTCAE criteria and logistic ordinal regression to understand the impact of PGx-guided prescribing on ADR intensity.
Incidence of clinically relevant adverse drug reactions (ADR) | 3 months
  Track the occurrence (incidence) of clinically relevant ADRs caused by the index or subsequent drugs as a binary outcome to preliminarily assess the safety of PGx-guided medication selection.
Serious adverse drug reactions | 3 months
  Focus on serious ADRs (frequency of ADRs) occurring within three months post-index drug administration to gain insights into the immediate safety impacts of PGx-guided versus standard care.
Self-Reported Adverse Drug Events (ADEs): | 3 months
  Collect data on all frequencies of self-reported ADEs, regardless of severity or drug-gene association, monthly over three months, providing a participant-centered view of drug tolerability.
Serious self reported adverse drug events (ADEs) | 3 months
  Track serious ADEs (frequency of ADEs) reported by participants, adding depth to the safety evaluation and focusing on participant-experienced impact
Dose Adjustments for Index Drug | 3 months
  Record the frequency of dose adjustments made for the index drug, capturing how PGx information influences pharmacotherapy adjustments.
Drug cessation due to adverse drug reactions (ADRs) | 3 months
  Monitor instances (frequency) of where the index drug is discontinued because of ADRs, offering a direct measure of drug tolerability under PGx-guided care.
Drug cessation due to lack of efficacy | 3 months
  Track discontinuations (frequency) of drugs due to lack of efficacy, providing a preliminary measure of the therapeutic effectiveness of PGx-guided prescribing.
14. Additional Prescribed Drugs During Follow-Up | 3 months
  Count additional drugs prescribed (frequency of additional drugs prescribed) during the follow-up period to gauge the potential broader impact of PGx testing on medication management complexity.
Changes in Drug Adherence | 3 months
  Evaluate changes in adherence scores from baseline to three months, exploring the influence of PGx testing on participant engagement and compliance. This will be assessed using the Medication Adherence Report Scale (MARS-5 questionnaire). Individual items will be scored 5 = never to 1 = always) i.e. high scores = high adherence. The total individual scores together to form a scale score (range = 5 to 25). Then an adjusted mean score is calculated by dividing the scale mean by the number of items in the scale (range 1-5).* The distribution of scores to see whether the scale should be dichotomised or left as a continuous scale. (In some data sets reported adherence is heavily positively skewed and in this case it might be advisable to dichotomise on the basis of the frequency distribution).
  *Point 3 is included to facilitate comparison across data sets where different versions of the MARS have been used (e.g. MARS-5: MARS-10 etc).
Participant Perspectives | 3 months
  Gather participants' perspectives on PGx testing through a survey administered at three months post-randomization, providing insights into participant experience and perceived value of PGx-guided care.

OTHER OUTCOMES:
Sub-group analysis- Age | 3 months
  Intervention effects on the primary and selected secondary outcomes will be compared between subgroups using interactions within regression models. Subgroups defined by the age of participants.
Sub-group analysis - Sex | 3 months
  Intervention effects on the primary and selected secondary outcomes will be compared between subgroups using interactions within regression models. Subgroups defined by the sex of participants.
Sub-group analysis- Scottish Index of Multiple Deprivation (SIMD) | 3 months
  Intervention effects on the primary and selected secondary outcomes will be compared between subgroups using interactions within regression models. Subgroups defined by the SIMD of participants.
Sub-group analysis- Ethnicity | 3 months
  Intervention effects on the primary and selected secondary outcomes will be compared between subgroups using interactions within regression models. Subgroups defined by the ethnicity of participants.
Sub-group analysis- Baseline polypharmacy burden | 3 months
  Intervention effects on the primary and selected secondary outcomes will be compared between subgroups using interactions within regression models.
  Subgroups defined by the baseline polypharmacy burden of participants.
Sub-group analysis- Consent type (participant/legal representative) | 3 months
  Intervention effects on the primary and selected secondary outcomes will be compared between subgroups using interactions within regression models. Subgroups defined by the consent type (participant/legal representative).

CONTACTS AND LOCATIONS:
Overall Officials: Sandosh Padmanabhan, MD PhD, Principal Investigator — University of Glasgow
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan for sharing individual participant data

REFERENCES:
- [Background] Swen JJ, van der Wouden CH, Manson LE, Abdullah-Koolmees H, Blagec K, Blagus T, Bohringer S, Cambon-Thomsen A, Cecchin E, Cheung KC, Deneer VH, Dupui M, Ingelman-Sundberg M, Jonsson S, Joefield-Roka C, Just KS, Karlsson MO, Konta L, Koopmann R, Kriek M, Lehr T, Mitropoulou C, Rial-Sebbag E, Rollinson V, Roncato R, Samwald M, Schaeffeler E, Skokou M, Schwab M, Steinberger D, Stingl JC, Tremmel R, Turner RM, van Rhenen MH, Davila Fajardo CL, Dolzan V, Patrinos GP, Pirmohamed M, Sunder-Plassmann G, Toffoli G, Guchelaar HJ; Ubiquitous Pharmacogenomics Consortium. A 12-gene pharmacogenetic panel to prevent adverse drug reactions: an open-label, multicentre, controlled, cluster-randomised crossover implementation study. Lancet. 2023 Feb 4;401(10374):347-356. doi: 10.1016/S0140-6736(22)01841-4. PMID 36739136
- [Background] Manson LE, van der Wouden CH, Swen JJ, Guchelaar HJ. The Ubiquitous Pharmacogenomics consortium: making effective treatment optimization accessible to every European citizen. Pharmacogenomics. 2017 Jul;18(11):1041-1045. doi: 10.2217/pgs-2017-0093. Epub 2017 Jul 7. No abstract available. PMID 28685652
- [Background] Samwald M, Xu H, Blagec K, Empey PE, Malone DC, Ahmed SM, Ryan P, Hofer S, Boyce RD. Incidence of Exposure of Patients in the United States to Multiple Drugs for Which Pharmacogenomic Guidelines Are Available. PLoS One. 2016 Oct 20;11(10):e0164972. doi: 10.1371/journal.pone.0164972. eCollection 2016. PMID 27764192
- [Background] Mallal S, Phillips E, Carosi G, Molina JM, Workman C, Tomazic J, Jagel-Guedes E, Rugina S, Kozyrev O, Cid JF, Hay P, Nolan D, Hughes S, Hughes A, Ryan S, Fitch N, Thorborn D, Benbow A; PREDICT-1 Study Team. HLA-B*5701 screening for hypersensitivity to abacavir. N Engl J Med. 2008 Feb 7;358(6):568-79. doi: 10.1056/NEJMoa0706135. PMID 18256392